CLINICAL TRIAL: NCT01798784
Title: Testing Behavioral Economic Interventions to Improve Statin Use and Reduce CVD Risk
Brief Title: Habit Formation for Adherence to Statin Use and LDL Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other); Rutgers University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AG043844-01 (NIH); 5R01AG043844 (NIH)
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Arm (No Intervention): Arm 1 will be the Control arm, in which participants receive an electronic pill container and are provided with daily reminders to take their medication but are not enrolled in the sweepstakes.
- Sweepstakes Incentive 1 (Experimental): Arm 2 will be a sweepstakes incentive arm where participants receive an electronic pill container and daily reminders to take their medication. In addition, this group is enrolled in a sweepstakes, in which participants may win money if they remember to take their medication.
  Interventions: Behavioral: Sweepstake Incentive 1
- Sweepstake Incentive 2 (Experimental): Arm 3 will be a sweepstake incentive arm where participants receive an electronic pill container and daily reminders to take their medication. In addition, this group is enrolled in a sweepstakes, in which monetary prizes may be awarded if participants take their medication prior to receiving a reminder.
  Interventions: Behavioral: Sweepstake Incentive 2
- Sweepstake Incentive 3 (Experimental): Arm 4 will be a sweepstake incentive arm where participants receive an electronic pill container and daily reminders to take their medication. In addition, this group is enrolled in a sweepstakes, in which each participant maintains an account that will accumulate money based on their medication adherence throughout the study.
  Interventions: Behavioral: Sweepstake Incentive 3

INTERVENTIONS:
Behavioral: Sweepstake Incentive 1 — Daily sweepstake conditional on daily medication adherence
  Arms: Sweepstakes Incentive 1
Behavioral: Sweepstake Incentive 2 — Daily sweepstake conditional on daily medication adherence
  Arms: Sweepstake Incentive 2
Behavioral: Sweepstake Incentive 3 — Daily sweepstake conditional on daily medication adherence
  Arms: Sweepstake Incentive 3

SUMMARY:
In a 4-arm, Randomized Control Trial among members of CVS Caremark or Penn Medicine Patients with suboptimal cholesterol control who are at high risk for CVD, the study investigators propose to test the effectiveness of different behavioral economic techniques in inducing habit formation for adherence to statin use and sustained reductions in LDL cholesterol after financial incentives are discontinued. Primary outcome is changes in LDL from enrollment to 12 months (6 months after cessation of financial incentives).

ELIGIBILITY:
Inclusion Criteria:

* Individuals at high risk of a cardiac event, specifically one of the following:
* Individuals with clinical CVD (defined as diagnosis with myocardial infarction, stroke, or peripheral vascular disease) with an LDL greater than or equal to 100 mg/dl ;
* Individuals with Diabetes (between the ages of 40-75) with an LDL greater than or equal to 100 mg/dl;
* Individuals without clinical CVD or diabetes with LDL greater than or equal to 100 mg/dl and estimated 10-year CVD risk 7.5%;
* Individuals without clinical CVD or diabetes with LDL cholesterol greater than or equal to 190 mg/dl A prescription filled for a statin medication within the last 12 months (derived from pharmacy records);
* Medication Possession Ratio (MPR) less than or equal to 80%
* Low medication adherence on self-report completed during enrollment

Exclusion Criteria:

* Less than 18 years old
* Contraindication to further statin use or have suffered side effects from statins, such as myopathy
* Will not or cannot give consent
* History of active or progressive liver disease or abnormal liver function tests on baseline screening when applicable
* Currently participating in another clinical trial with related aims
* Co-morbidities likely to lead to death within a short-period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in LDL from baseline to 12 months | 12 months

SECONDARY OUTCOMES:
Statin Adherence 6 months after active phase of intervention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; Iwan Barankay, PhD, Principal Investigator — University of Pennsylvania; Peter Reese, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Barankay I, Reese PP, Putt ME, Russell LB, Phillips C, Pagnotti D, Chadha S, Oyekanmi KO, Yan J, Zhu J, Volpp KG, Clapp JT. Qualitative Exploration of Barriers to Statin Adherence and Lipid Control: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e219211. doi: 10.1001/jamanetworkopen.2021.9211. PMID 33944923
- [Derived] Russell LB, Norton LA, Pagnotti D, Sevinc C, Anderson S, Finnerty Bigelow D, Iannotte LG, Josephs M, McGilloway R, Barankay I, Putt ME, Reese PP, Asch DA, Goldberg LR, Mehta SJ, Tanna MS, Troxel AB, Volpp KG. Using Clinical Trial Data to Estimate the Costs of Behavioral Interventions for Potential Adopters: A Guide for Trialists. Med Decis Making. 2021 Jan;41(1):9-20. doi: 10.1177/0272989X20973160. Epub 2020 Nov 20. PMID 33218296
- [Derived] Barankay I, Reese PP, Putt ME, Russell LB, Loewenstein G, Pagnotti D, Yan J, Zhu J, McGilloway R, Brennan T, Finnerty D, Hoffer K, Chadha S, Volpp KG. Effect of Patient Financial Incentives on Statin Adherence and Lipid Control: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2019429. doi: 10.1001/jamanetworkopen.2020.19429. PMID 33034639
- [Derived] Putt ME, Reese PP, Volpp KG, Russell LB, Loewenstein G, Yan J, Pagnotti D, McGilloway R, Brennen T, Finnerty D, Hoffer K, Chadha S, Barankay I. The Habit Formation trial of behavioral economic interventions to improve statin use and reduce the risk of cardiovascular disease: Rationale, design and methodologies. Clin Trials. 2019 Aug;16(4):399-409. doi: 10.1177/1740774519846852. Epub 2019 May 31. PMID 31148473